CLINICAL TRIAL: NCT05093699
Title: Dual-plane Ultrasound Imaging During Vascular Access Procedures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Robert (Bobby) J. Anderson, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 21-007039
Record Dates: First submitted 2021-10-13; First posted 2021-10-26 (Actual); Results first posted 2024-07-31 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-05

CONDITIONS: Vascular Access Complication

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Control Group (Active Comparator): Arterial line placement via standard mechanism; utilization of a single-plane ultrasound probe
  Interventions: Device: Ultrasound probe
- Butterfly iQ+ ultrasound probe (Experimental): Arterial line placement utilizing dual-plane, Butterfly iQ+ ultrasound probe
  Interventions: Device: Butterfly iQ+ ultrasound probe

INTERVENTIONS:
Device: Butterfly iQ+ ultrasound probe — Diagnostic ultrasound probe on-market (FDA approved) capable of dual-plane viewing
  Arms: Butterfly iQ+ ultrasound probe
Device: Ultrasound probe — Standard single-view ultrasound probe
  Arms: Control Group

SUMMARY:
Researchers are evaluating the clinical efficiency of utilization of a dual-plane simultaneous view ultrasound probe (Butterfly iQ+; Butterfly Network, Inc.) during arterial catheter placement in the operating room

ELIGIBILITY:
Inclusion criteria

* Patient: Elective surgical patients requiring non-emergent ultrasound-guided radial arterial catheter placement
* Providers: Anesthesia providers to include trainees, certified registered nurse anesthetists (CRNA) and attending anesthesia providers.

Exclusion Criteria

* Patient
* Pregnant
* Patients in a moribund state or palliative care only
* Vulnerable patients (i.e. Severe mental handicap, non-decisional)
* History of peripheral arterial disease
* Placement of arterial catheter without ultrasound guidance
* Provider: Medical students or CRNA students.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2024-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Anderson, APRN, CNP, DNP, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic - Clinical Trials — https://www.mayo.edu/research/clinical-trials/cls-20530185

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control Group | Butterfly iQ+ Ultrasound Probe
Started | 50 | 48
Completed | 50 | 48
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group | Butterfly iQ+ Ultrasound Probe | Total
Number analyzed (Participants) | 50 | 48 | 98
Age, Continuous [Mean (Full Range); unit: years] | 50 [18 to 85] | 50 [18 to 85] | 50 [18 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 24 | 49
  Male | 25 | 24 | 49
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 50 | 48 | 98
Analyzed [Count of Participants; unit: Participants] | 50 | 48 | 98

OUTCOME MEASURES:

1. Primary Outcome: Time to Successful First Stick in Minutes
Description: Number of first-stick success rate of ultrasound-guided peripheral arterial catheter placement
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Control Group | Butterfly iQ+ Ultrasound Probe
Number analyzed (Participants) | 50 | 48
minutes | 4.56 (3.95) | 6.24 (5.36)

2. Secondary Outcome: Number of Attempts for Successful Cannulation
Description: Number of attempts to achieved successful arterial catheter cannulation; attempt will be defined as a single insertion of the needle into the skin.
Time Frame: Arterial line placement episode for surgery
Measure: Number; unit: Successful arterial line placement
Arm/Group | Control Group | Butterfly iQ+ Ultrasound Probe
Number analyzed (Participants) | 50 | 48
Successful arterial line placement | 48 | 39

3. Secondary Outcome: Amount of Time Required for Successful Arterial Catheter Cannulation
Description: Amount of time measured in minutes for successful arterial catheter cannulation
Time Frame: Baseline
Measure: Mean (Full Range); unit: minutes
Arm/Group | Control Group | Butterfly iQ+ Ultrasound Probe
Number analyzed (Participants) | 50 | 48
minutes | 4.56 [0.20 to 18.01] | 6.24 [0.42 to 22.54]

4. Secondary Outcome: Number of Failed Attempts for Cannulation
Description: Number of failed attempts leading to unsuccessful arterial catheter cannulation
Time Frame: Baseline
Measure: Number; unit: number of failed attempts
Arm/Group | Control Group | Butterfly iQ+ Ultrasound Probe
Number analyzed (Participants) | 50 | 48
number of failed attempts | 2 | 9

ADVERSE EVENTS:
Time Frame: Total study - 6 months
Arm/Group | Control Group | Butterfly iQ+ Ultrasound Probe
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/48
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/48
Other Adverse Events (participants affected / at risk) | 0/50 | 0/48

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2021-11-02): https://cdn.clinicaltrials.gov/large-docs/99/NCT05093699/Prot_002.pdf
  • Statistical Analysis Plan (2023-09-01): https://cdn.clinicaltrials.gov/large-docs/99/NCT05093699/SAP_003.pdf
  • Informed Consent Form (2021-07-12): https://cdn.clinicaltrials.gov/large-docs/99/NCT05093699/ICF_001.pdf